CLINICAL TRIAL: NCT06020742
Title: Automitochondrial Transplantation Improves Live Birth in Elderly Patients With Low Prognosis After Repeated IVF Failure
Acronym: ACTILB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Han Hongjing, chief physician, Peking University People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDL2022-25
Record Dates: First submitted 2023-08-03; First posted 2023-09-01 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Infertility, Female; Mitochondrial; Elderly; Assisted Reproductive Technique
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MT transfer (Experimental)
  Interventions: Procedure: Autologous USC mitochondrial oocyte transplantation

INTERVENTIONS:
Procedure: Autologous USC mitochondrial oocyte transplantation — Mitochondria are isolated from urine derived stem cells from fresh middle urine of the subjects, and injected into the cytoplasm of mature oocytes together with sperm

SUMMARY:
The goal to this clinical trial is to study the effectiveness and safety of automitochondrial transplantation of urine derived stem cells(USCs) in in elderly patients with low prognosis after repeated IVF failure. The main questions it aims to answer are:

(1）test the effectiveness and safety of automitochondrial transplantation of urine derived stem cells (2) establish intracytoplasmic sperm injection(ICSI) mitochondrial transplantation platform Participants will be asked to:1)urine collections to further culture of autologous USCs 2)ovarian stimulation、trigger eggs、ICSI with autologous mitochondria 3）embryo transfer 4)accept pregnancy follow-up at given point

ELIGIBILITY:
Inclusion Criteria:

1. 1) At least 35 years old
2. 2) Repeated IVF failure: more than or equal to 2 egg retrieval with poor embryo quality, no transplanted embryos or failed embryo transfer (more than or equal to 4 embryos)
3. 3) Egg number ≤9
4. 4) Participate voluntarily and sign informed consent.

Exclusion Criteria:

1: Infertility caused by severe oligospermia, severe intrauterine adhesions, genital tract malformations, thyroid dysfunction and other endocrine, immune system, tumor and genetic diseases

Min Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
live birth rate | 1year after embryo transfer
  Live birth rate per embryo transfer cycle (defined as live delivery after ≧28 weeks)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's hospital, Beijing, Beijing Municipality, China